CLINICAL TRIAL: NCT02794051
Title: Implementation of a Transdiagnostic Group Intervention for Children With Behavior Problems Within a Pediatric Outpatient Setting
Brief Title: Transdiagnostic Group Intervention for Children With Behavior Problems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Children's Hospital Colorado (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-0275
Record Dates: First submitted 2016-05-17; First posted 2016-06-08 (Estimated); Last update posted 2016-09-29 (Estimated); Status verified 2016-09

CONDITIONS: Behavioral Symptoms; Emotional Disturbances
MeSH Terms: conditions — Behavioral Symptoms; Affective Symptoms | interventions — Psychotherapy, Group

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Unified Protocol for Children (Experimental): Child participants with behavior problems between the ages of 8-12 and their caregivers will participate in a transdiagnostic group therapy protocol.
  Interventions: Behavioral: Group Therapy

INTERVENTIONS:
Behavioral: Group Therapy — Participating children and their caregivers will attend 90-minute weekly group therapy sessions for 10 consecutive weeks.

SUMMARY:
This study fills a notable gap in the transdiagnostic literature by evaluating whether an evidence-based transdiagnostic treatment for emotional disorders such as the Unified Protocol for Children (UP-C) is effective for treating childhood behavior problems.

DETAILED DESCRIPTION:
By participating in the study, child participants will learn emotion regulation skills and have opportunities to interact and practice skills with other children who have similar problems. In addition, parent participants will learn effective parenting skills, including appropriate limit-setting, use of praise and consequences, and empathy, that may help them effectively navigate the challenges of caring for a child with behavior concerns (1). Parents will also have the opportunity to interact with other parents who face similar challenges, providing validation and support. Upon completion of the study, investigators plan to share these findings at professional conferences and submit manuscripts to peer-reviewed journals. Collectively, this study will add to the literature in the pediatric mental health field and may also serve as a model for other outpatient clinics regarding implementation and provision of a transdiagnostic approach to treat children with behavior problems. Thus, the main goals of the current study are to examine the effectiveness of the UP-C group treatment in reducing childhood behavior problems, evaluate parents' satisfaction with this treatment, and determine the feasibility of implementing this treatment in a pediatric outpatient setting.

ELIGIBILITY:
Inclusion Criteria:

* Ages 8 - 12 years
* English speaking
* Primary Behavior Disorder
* At least 1 English-speaking parent/legal guardian who can provide informed consent for the child
* Parent/Legal Guardian must agree to participate in the Trial

Exclusion Criteria:

* Child is: a ward of the state
* has active suicidal ideation
* has homicidal ideation
* has self-harm behaviors
* has an intellectual disability
* has a pervasive developmental disability or significant developmental delay
* has an active substance use disorder
* is currently participating in individual or group psychotherapy, or
* has participated in therapy within the past year
* has a sibling that is also enrolled in the study
* Parents/Legal Guardians that:

  1. are unwilling to participate in the study
  2. are non-English speaking
  3. have an intellectual disability
  4. have a pervasive developmental disability or
  5. a significant developmental delay
  6. do not have legal custody of the child participant
  7. do not reside in the same home as the child participant

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 8 (Actual)
Dates: Start 2016-05; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Change in rates of noncompliance, tantruming, and parenting practices on the Home Record Card | 12 weeks - Measured daily from baseline to post-treatment
  Chart for recording events of noncompliance, tantrums, and parenting practices.

SECONDARY OUTCOMES:
Change in pre- vs. post-treatment scores on the Transdiagnostic Questionnaires for Parent and Child | 10 weeks - Measured at Week 1 (pre-treatment) and at Week 10 (post-treatment)
  Measures several transdiagnostic mechanisms including child emotional and behavioral symptoms, sleeping difficulties, and parenting practices.
Change in pre- vs. post-treatment scores on the Eyberg Child Behavior Inventory | 10 weeks - Measured at Week 1 (pre-treatment) and at Week 10 (post-treatment)
  Measures intensity of behavior related problems and degree to which these behaviors are viewed as problematic by parents.
Change in pre- vs. post-treatment scores on the Achenbach Rating Scales (Child Behavior Checklist and Youth Self-Report) | 10 weeks - Measured at Week 1 (pre-treatment) and at Week 10 (post-treatment)
  Measures parent and child report of the presence of child behavior and emotional problems
Change in pre- vs. post-treatment scores on the Alabama Parenting Questionnaire | 10 weeks - Measured at Week 1 (pre-treatment) and at Week 10 (post-treatment)
  Measures five dimensions of parenting: positive involvement, supervision, positive discipline techniques, consistency in disciplining, and use of corporal punishment.
Parents' satisfaction with treatment, as measured by the Family Satisfaction Survey | 10 weeks - Measured at weeks 3, 7, and 10.
  To assess parents' satisfaction with their participation in the UP-C intervention.
Treatment feasibility, as measured by the Family Satisfaction Survey and attendance rates | 10 weeks
  To evaluate parents' opinions about whether participation in a 10-week therapy group treatment is feasible and whether the interventions taught are feasible.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Malmberg, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
Single subject design data

REFERENCES:
- [Background] Ehrenreich-May et al., 2012